CLINICAL TRIAL: NCT05612724
Title: Rutgers Pilot for Pragmatic Return to Effective Dental Infection Control Through Triage and Testing (PREDICT)- Patient POC Test
Brief Title: Rutgers Pilot for PREDICT- Patient POC Test
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Principal Investigator, Cecile A. Feldman, DMD, Professor, Rutgers, The State University of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro2020002998; X01DE030407 (Other: NIDCR)
Record Dates: First submitted 2022-10-31; First posted 2022-11-10 (Actual); Results first posted 2024-03-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: SARS CoV 2 Infection
Keywords: Screening; Point-of-care testing; Asymptomatic patients; Perception of safety; Feasibility
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Pilot study to assess feasibility of testing asymptomatic dental patients for SARS-CoV-2 antigen using Rapid Antigen point-of-care testing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- SARS-CoV-2 testing (Other): There is only one arm in this study- the study is a non-randomized pilot. All the subjects will be tested for SARS CoV 2 viral Antigen as described.
  Interventions: Device: Testing for SARS CoV2 Antigen

INTERVENTIONS:
Device: Testing for SARS CoV2 Antigen — Device: Testing for SARS CoV2 Antigen Antigen testing: Rapid Antigen testing (Point-of-care)

SUMMARY:
A pilot study was initiated to assess feasibility of testing asymptomatic dental patients presenting to the Oral Medicine Clinic at Rutgers School of Dental Medicine for SARS-CoV-2 viral antigen using a point-of-care (POC) Rapid Antigen test.

14 subjects with upcoming appointment at the Oral Medicine clinic, Rutgers School of Dental Medicine, with no history of documented COVID-19 infection or viral exposure, were enrolled in a study that interrogated patients' perceptions of safety and feedback regarding their testing experience. All 14 patients expressed initial interest, however, 10 patients completed informed consent and completed study procedures.

Institutional Clinical Laboratory Improvement Amendments (CLIA) certification of waiver was obtained prior to conducting the study. Communicable Diseases Reporting and Surveillance System (CDRSS) registration and training were completed to enable reporting results of the POC test.

DETAILED DESCRIPTION:
A pilot study was initiated to assess feasibility of testing asymptomatic dental patients presenting to the Oral Medicine Clinic at Rutgers School of Dental Medicine for SARS-CoV-2 viral antigen using a point-of-care (POC) Rapid Antigen test.

14 subjects with upcoming appointment at the Oral Medicine clinic, Rutgers School of Dental Medicine, with no history of documented COVID-19 infection or viral exposure, were enrolled in a study that interrogated patients' perceptions of safety and feedback regarding their testing experience. All 14 patients expressed initial interest, however, 10 patients completed informed consent and completed study procedures on their appointments, the remaining 4 patients did not present for their appointment.

Following initial interest in participation over the phone, the subjects completed a pre-visit survey prior to their upcoming appointment. The day prior to their visit, a phone triage was completed and repeated as they checked in for their appointment. A nasal sample was collected and processed using the FDA EUA authorized Rapid Antigen Test BD Veritor Plus Analyzer, BD Sciences. An end-of-study survey was collected to assess patients' feedback about their experience and their perception of safety.

ELIGIBILITY:
Inclusion Criteria:

* Dental Patients with upcoming appointment at the Oral Medicine Clinic at Rutgers School of Dental Medicine

Exclusion Criteria:

* Patients previously participating in the study
* Patients unwilling to have their de-identified data made available to researchers

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-12-30 (Actual); Primary Completion 2021-01-20 (Actual); Study Completion 2022-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cecile A Feldman, Principal Investigator — Rutgers School of Dental Medicine
Locations (1):
- Rutgers School of Dental Medicine, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
D: No If the COVID test results show that a participant is positive for COVID-19, the study staff will tell the participant the results. The study staff will be required to give the participant's name to the state's Department of Public Health if the participant tests positive because this is the law.
  At the end of the study, de-identified data will be provided to the National Coordinating Center.

REFERENCES:
- [Background] 1. American Dental Association COVID-19 Toolkit - Update to Office Procedures During COVID-19. https://www.ada.org/-/media/project/ada-organization/ada/ada-org/files/resources/coronavirus/update_to_office_procedures_during_covid19.pdf accessed on November 11, 2021.
- [Background] Estrich CG, Mikkelsen M, Morrissey R, Geisinger ML, Ioannidou E, Vujicic M, Araujo MWB. Estimating COVID-19 prevalence and infection control practices among US dentists. J Am Dent Assoc. 2020 Nov;151(11):815-824. doi: 10.1016/j.adaj.2020.09.005. PMID 33071007
- [Background] Shirazi S, Stanford CM, Cooper LF. Testing for COVID-19 in dental offices: Mechanism of action, application, and interpretation of laboratory and point-of-care screening tests. J Am Dent Assoc. 2021 Jul;152(7):514-525.e8. doi: 10.1016/j.adaj.2021.04.019. Epub 2021 May 4. PMID 34176567

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 14 asymptomatic dental patients with upcoming appointments at the Oral Medicine Clinic, Rutgers School of Dental Medicine, were enrolled. Study participation took place in between December 2020 and January 2021.
Period: Overall Study
Arm/Group | SARS-CoV-2 Testing
Started | 14
Completed | 10
Not Completed | 4
Not completed — Lost to Follow-up | 4

BASELINE CHARACTERISTICS:
Arm/Group | SARS-CoV-2 Testing
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.9 (17.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 3
  More than one race | 1
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Patient Willingness to Follow Through With the Study Surveys, Triage and Testing
Description: Percentage of 14 patients who complete the study
Time Frame: Through study completion, an average of 21 days
Population: 14 patients enrolled in the study. The percentage of 14 patients who completed the study is tabulated
Measure: Number; unit: percentage of participants
Arm/Group | SARS-CoV-2 Testing
Number analyzed (Participants) | 14
percentage of participants | 71.42

2. Primary Outcome: Patient Test Completion
Description: Percentage of 14 patients with completed SARS-CoV-2 testing
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | SARS-CoV-2 Testing
Number analyzed (Participants) | 14
Participants | 10

3. Primary Outcome: Patient Ease of Complying With Protocol
Description: Number of participants indicating that it was easy to complete the surveys
Time Frame: Day 21
Measure: Count of Participants; unit: Participants
Arm/Group | SARS-CoV-2 Testing
Number analyzed (Participants) | 10
Participants | 10

4. Primary Outcome: Percentage of Surveys Completed by Patients
Description: Percentage of patients with completed pre-visit, triage and post-visit surveys completed
Time Frame: Through study completion (21 days)
Measure: Count of Participants; unit: Participants
Arm/Group | SARS-CoV-2 Testing
Number analyzed (Participants) | 14
Participants | 10

ADVERSE EVENTS:
Time Frame: From signing initial consent to completion of study- 21 days
Description: This study involved a nasal swab and a survey
Arm/Group | SARS-CoV-2 Testing
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-10-17): https://cdn.clinicaltrials.gov/large-docs/24/NCT05612724/Prot_SAP_000.pdf
  • Informed Consent Form (2020-12-15): https://cdn.clinicaltrials.gov/large-docs/24/NCT05612724/ICF_002.pdf